CLINICAL TRIAL: NCT04262596
Title: Effectiveness of an Interactive Consulting System to Enhance Patients' Decision-making: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2020KYPJ002
Record Dates: First submitted 2020-01-23; First posted 2020-02-10 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Age-related Cataract

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Consulting System (Experimental): The AI system adheres to the AHRQ SHARE approach (https://www.ahrq.gov/health-literacy/professional-training/shared-decision/tools/factsheet.html) for shared decision-making, which involves evaluating healthcare options, weighing pros and cons, and assessing potential risks while allowing patients to express their preferences.
  Interventions: Other: Interactive Consulting System
- Traditional decision aid brochure (Active Comparator): A traditional patient decision aid brochure that includes provide standard general information, quantitative risk information on the possible outcomes of cataract surgery and value clarification exercise.
  Interventions: Other: A traditional patient decision aid brochure

INTERVENTIONS:
Other: Interactive Consulting System — Potential participants use the Interactive Consulting System on a mobile application with information about cataract surgery choice, and outcome data will be gathered using standardized questions in a structured interview after 2 weeks.
  Arms: Interactive Consulting System
Other: A traditional patient decision aid brochure — Potential participants receive a traditional patient decision aid brochure with information about cataract surgery choice, and outcome data will be gathered using standardized questions in a structured interview after 2 weeks.
  Arms: Traditional decision aid brochure

SUMMARY:
To compare the effectiveness of an interactive mobile chatbot and traditional decision aid booklets to enhance informed decisions made by cataract patients. The chatbot was built based on large language models, and could generate ChatGPT-level responses.

DETAILED DESCRIPTION:
Cataract surgery is the only way to treat age-related cataract. For patients at early or moderate stages, cataract surgery is an elective surgery without objective indications. Therefore, patients are uaually not aware whether they should receive the surgery or not. In clinical practice, traditional Patient Decision Aids (PDA) booklets are used to provide health education to patients. However, PDAs lack real-time interaction with patients, and are unable to answer the new questions raised. Patients still have doubts about whether they should receive cataract surgery or not. In this study, the investigators aim to assess the effectiveness of an interactive Q&A mobile application based on natural language processing technology to enhance informed decisions made by cataract patients.

ELIGIBILITY:
Inclusion Criteria

1. Individuals aged 50-80, living in the designated research area for more than 6 months;
2. Primary diagnosis of cataract and have not undergone cataract surgery;
3. Ownership of a smartphone/tablet capable of using the study app and the ability to smoothly type in chat content
4. Willing to participate in the research and provide informed content.

Exclusion Criteria

1. Blindness in both eyes (manifesting as a distant vision less than 3/60);
2. Eye, hearing, or mental disorders that hinder reading or telephone interviews;
3. Permanent vision loss due to eye diseases other than cataracts, which cannot be corrected by cataract surgery;
4. Contraindications for cataract surgery.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Informed choice about cataract surgery (the proportion of participants who make an informed choice，which is defined as a good knowledge score and an intention that is consistent with their attitude score) | 2 weeks post intervention
  Informed choice is an aggregated measure of multiple measurements, including:
  1. Knowledge (a 12-item questionnaire that assesses conceptual knowledge of cataract and cataract surgery). Questions with right answers will earn 1 point otherwise 0 point. Each participant may get 12 points maximally and 0 point minimally.
  2. Attitudes (6 items, with 5 responses for each. Each response will earn 0-4 points respectively);
  3. Intentions (single item with 5 responses. Each response will earn 0-4 points respectively).
  Higher scores indicate a better knowledge on informed choice of cataract surgery.

SECONDARY OUTCOMES:
Decisional conflict | 2 weeks post intervention
  Decisional conflict will be assessed using a 16-item Decisional Conflict Scale. Each item has 5 responses. Each response will earn 0-4 points respectively. Lower scores indicate a stronger ability to decide wheter or not receiving a cataract surgery.
Decisional confidence | 2 weeks post intervention
  Decisional confidence will be assessed using a 11-item Decision Self Efficacy Scale. Each item has 5 responses. Each response will earn 0-4 points respectively. Higher scores indicate the paricipant is more confident about his/her decision.
Time perspective | 2 weeks post intervention
  This will be assessed using a 4-item short form of the Consideration of Future Consequences Scale, with five response categories ranging from strongly agree (4 points) to strongly disagree (0 point). Higher scores indicate more consideration of future consequences by the participants.
Anticipated regret | 2 weeks post intervention
  Two items from a validated scale will measure anticipated regret about having cataract surgery (action regret, 4 points) and about not having cataract (inaction regret, 0 point). Higher scores indicate higher probability of anticipated regret after the surgery.
Cataract worry | 2 weeks post intervention
  A validated single item will measure participants' level of worry about progression of cataract, using four verbal response categories ranging from not worried at all to very worried. There are five response categories ranging from strongly agree (3 points) to strongly disagree (0 point). Higher scores indicate more worried about the disease status.
Cataract anxiety | 2 weeks post intervention
  Anxiety will be measured with a six-item short form.A validated single item will measure participants' level of worry about progression of cataract, using four verbal response categories ranging from not worried at all to very worried. Each question has five response categories ranging from strongly agree (3 points) to strongly disagree (0 point). Higher scores indicate more anxious about the disease status.
Perceived importance of surgical benefit/harms | 2 weeks post intervention
  Purpose-developed items will be used to ask participants about their personal perceptions of the importance of specific outcomes in their decision-making about cataract surgery. The questionare contains 2 items with 5 responses. Each response will earn 0-4 points respectively). Higher scores indicate a better knowledge on the understanding of importance of surgical benefit/harms.
Perceived importance of surgical benefit/harms | Time Frame: 2 weeks post intervention
  Purpose-developed items will be used to ask participants about their personal perceptions of the importance of specific outcomes in their decision-making about cataract surgery. The questionnaire contains 2 items, each with 5 responses14. Each response will earn 0-4 points respectively). Higher scores indicate a better knowledge on the understanding of importance of surgical benefit/harms.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfeng Zheng, Principal Investigator — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No